CLINICAL TRIAL: NCT00630266
Title: Clinical Evaluation of Acorn CorCap Cardiac Support Device Concomitant to MVR - A Confirmatory Trial
Brief Title: Confirmation Trial of the Acorn CorCap Cardiac Support Device (CSD) at the Same Time as Mitral Valve Repair
Acronym: MVR + CorCap
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acorn Cardiovascular, Inc. (Industry)
Responsible Party: Steve Anderson, President, Acorn Cardiovascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 47-1389
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Heart Failure
Keywords: Heart failure; left ventricular dilation; mitral valve repair; mitral valve replacement
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CorCap CSD — The surgical procedure includes implantation of the CorCap CSD with concommitant mitral valve surgery through a sternotomy.

SUMMARY:
The purpose of this study to evaluate patients when they have an Acorn CorCapTM Cardiac Support Device (CSD) placed around their heart for the treatment of heart failure at the same time as their mitral valve surgery.

The CorCapTM CSD is intended to support the heart, potentially preventing further dilation that is associated with progressive heart failure, thereby potentially preserving or improving heart function.

DETAILED DESCRIPTION:
The Acorn CorCap Cardiac Support Device (CSD) is a new therapy for the treatment of heart failure that is designed to reduce left ventricular dilation, which is one of the most important pathophysiological mechanisms underlying the clinical syndrome of heart failure. The Acorn CorCap CSD is intended to reduce wall stress and support the heart, in order to prevent further dilation that is associated with progressive heart failure. It is designed to result in reduced left ventricular size and improve left ventricluar function, which should result in improved patient functional status.

The purpose of the study is to provide confirmatory data to demonstrate an improved benefit-risk profile in support of a Pre-Market Approval (PMA) application for the Acorn CorCap CSD when placed concomitant to Mitral Valve Repair/Replacement (MVR).

The primary efficacy objective is to evaluate patient functional status after 6 months of follow-up. The safety endpoint is perioperative (30 day) mortality.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy of either ischemic or non-ischemic origin
* Patients must be on stable, optimally uptitrated medical therapy recommended according to current guidelines as standard of care of heart failure therapy in the United States. This minimally includes:

  1. Angiotensin-converting enzyme inhibitors (ACE) or alternate if ACE not tolerated for greater than or equal to 1 month prior to enrollment (not required for patients with a mitral valve anomaly that is not likely to respond to medication and requires surgical intervention).
  2. Treatment with a beta-blocker, unless intolerant, for greater than or equal to 3 months prior to enrollment (not required for patients with a mitral valve anomaly that is not likely to respond to medication and requires surgical intervention).
  3. Diuretic at least "prn" (as occasion requires).
  4. Cardiac medications unchanged for greater than or equal to 1 month except for diuretic adjustments (not required for patients with a mitral valve anomaly that is not likely to respond to medications and requires surgical intervention).
* Adult (18 to 80 years).
* Indexed left ventricular end diastolic dimension (LVEDDi)between 30 mm/m2 and 40 mm/m2 as determined by transthoracic echocardiography.
* Mitral regurgitation (MR) greater than or equal to 2+ and scheduled for mitral valve repair or replacement. Concomitant tricuspid valve repair or replacement (TVR) and/or atrial fibrillation ablation procedures will be permitted.
* Left ventricular ejection fraction (LVEF) less than or equal to 45 percent via transthoracic echocardiography, cardiac catheterization, radionuclide scan, or magnetic resonance imaging
* New York Heart Association Functional Class (NYHA) II, III or IV
* Geographically available for follow-up
* Signed Informed Consent

Exclusion Criteria:

* Inability to reach maximal effort CPX test as defined by the CPX Core Lab
* Planned cardiac surgical procedure other than MVR
* Hypertrophic obstructive cardiomyopathy.
* Significant cardiomegaly, which is estimated to exceed the largest available size of CorCap CSD.
* Expectation of existing cardiothoracic adhesions that would cause an inability to gain complete circumferential access to the heart.
* Existing patent CABG.
* Candidates for surgical revascularization as determined by an angiogram. Patients with ischemic heart disease who have not had an angiogram within the past 3 years and in whom lesions amenable to revascularization cannot be excluded should have a repeat angiogram.
* Any condition considered a contraindication for extracorporeal circulation.
* Use of Intra aortic Balloon Pump (IABP), intravenous inotropic or vasoactive agents within 30 days prior to enrollment. Pre-operative hemodynamic optimization with IABP, IV inotropes or vasoactive agents may be permitted if it is scheduled to occur within 48 hours of planned index surgery.
* Current or anticipated need for left ventricular assist device (LVAD) or cardiac replacement device.
* Anticipated need for heart transplant within the next two years.
* Acute myocardial infarction (AMI), unstable angina, or cerebral vascular accident (CVA) or Transient Ischemic Attack (TIA) within past 3 months.
* Percutaneous coronary intervention (PCI) or transmyocardial laser revascularization (TMR or PMR) within the past 3 months.
* Presence of arrhythmias causing hemodynamic instability, history of resuscitated sudden death without subsequent treatment with implantable defibrillator or amiodarone, or atrial fibrillation with a ventricular rate greater than 100 bpm on medication.
* Co-morbid condition that reduces life expectancy to less than 1 year.
* Active infection.
* Pregnancy at the time of enrollment. (Women of child bearing potential must have a negative serum pregnancy test within two weeks prior to enrollment, or be using hormonal contraceptives or intrauterine devices.)
* Enrolled in another investigational study that would confound interpretation of trial results.
* Patients who participated as control patients in the previous CorCap PMA randomized trial.
* Unable to comply with protocol-required follow-up (as judged by primary investigator or referring cardiologist).
* Late stage heart failure with increased surgical risk as defined by the presence of four or more of the following:

  1. LVEDD greater than 80 mm/m2
  2. Resting systolic blood pressure (BP) less than or equal to 80 mm Hg (on clinical exam)
  3. Atrial fibrillation at time of enrollment or paced rhythm with underlying atrial fibrillation
  4. Heart failure greater than or equal to 8 years
  5. 6 minute walk less than or equal to 350 meters (1148 feet)
  6. POV2 less than or equal to 13 ml/kg/min (CPX test)
  7. Exercise induced increase in systolic BP less than 10 percent (CPX test)
  8. Previous cardiac surgery
  9. BUN greater than 100 mg/dl
  10. Cachexia (clinical impression)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient functional status as evaluated using the Minnesota Living with Heart Failure questionnaire | 6 month follow-up
Change in maximal exercise tolerance evaluated using cardiopulmonary exercise (CPX) testing (peak VO2 exercise test) | 6 Month follow-up
Change in sub-maximal exercise tolerance as evaluated using the Six Minute Walk test. | 6 months
Number of patients who have died (all-cause) or had a re-hospitalization due to heart failure. | 6 months
Peri-operative mortality, death occuring within 30 days of baseline surgery. | 30 days

SECONDARY OUTCOMES:
Rate of death and SAEs overall and for each specific type of event | 6 months
Change in patient functional status as evaluated using the Minnesota Living with Heart Failure Questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven F Bolling, MD, Principal Investigator — University of Michigan; Michael A Acker, MD, Principal Investigator — Hospital of the University of Pennsylvania, Cardiovascular Medicine; Penn-Presbyterian Medical Center; Mario Pompili, MD, Principal Investigator — Kaiser Permanente Northern California Heart Transplant Program; James Wudel, MD, Principal Investigator — Nebraska Heart Institute; Randall Starling, MD, Principal Investigator — The Cleveland Clinic; Mark J Zucker, MD, JD, Principal Investigator — Newark Beth Israel; Renzo Cecere, MD, Principal Investigator — Royal Victoria Hospital, McGill University; Pat Pappas, MD, Principal Investigator — advocate christ medical center; Robert Brewer, MD, Principal Investigator — Henry Ford Hospital; Jeff Cope, MD, Principal Investigator — Lancaster General Hospital; Edward Raines, MD, Principal Investigator — BryanLGH Medical Center
Locations (12):
- United States (11):
  - Kaiser Permanente Northern California Heart Transplant Program, Santa Clara, California
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - BryanLGH Medical Center, Lincoln, Nebraska
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Newark Beth Israel, Newark, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - PENN-Presbyterian Medical Center, Philadelphia, Pennsylvania
- Royal Victoria Hospital, McGill University, Montreal, Quebec, Canada